CLINICAL TRIAL: NCT03346174
Title: Influence of Assisted Autogenic Drainage (AAD) and Bouncing Combined With Assisted Autogenic Drainage (BAAD) on Acid and Non-acid Gastro-oesophageal Reflux (GOR) in Infants < 1 Year
Brief Title: Influence of Airway Clearance Techniques on GOR in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Filip Van Ginderdeuren, Prof. Dr., Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FVG004
Record Dates: First submitted 2017-11-09; First posted 2017-11-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Gastro-oesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data will be analyzed by an experienced paediatric gastro-enterologist, blinded to the different treatment modalities
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AAD (Experimental): AAD is an airway clearance technique for infants based upon the principles of autogenic drainage. By modulating manually the functional breathing level within the vital capacity, optimal airflow will be obtained at the targeted airway generations, where secretions have been identified. A gentle increase of manual pressure on the chest during each inspiration is performed to guide the breathing of the patient towards the desired lung volume level. During expiration the breathing movement of the patient is followed gently.
  Interventions: Other: AAD
- BAAD (Experimental): AAD is an airway clearance technique for infants based upon the principles of autogenic drainage .AAD sometimes leads to crying or resistance against therapy.Bouncing (at low amplitude:6-8 cm) in a stable upright position is a gentle up-and-down movement on a physio ball. It is not an ACT, but used to maximize the relaxation of the infant, avoiding resistance against or crying during treatment. Due to the relaxing effect of bouncing, infants appear to tolerate better AAD, increasing the effectiveness of the treatment.
  Interventions: Other: BAAD

INTERVENTIONS:
Other: AAD — In this controlled trial with intra-subject design infants will be studied using multichannel intraluminal impedance pH (pH-MII) monitoring , during which they receive one 20 min session of AAD . The number of reflux episodes (RE) is the outcome measure. The results obtained during and 20 min after the intervention will be compared to a period of 20 min before treatment ( control ).
  Arms: AAD
Other: BAAD — In this controlled trial with intra-subject design infants will be studied using multichannel intraluminal impedance pH (pH-MII) monitoring , during which they receive one 20 min session of BAAD . The number of reflux episodes (RE) is the outcome measure. The results obtained during and 20 min after the intervention will be compared to a period of 20 min before treatment ( control ).
  Arms: BAAD

SUMMARY:
The purpose of this study is to determine whether Assisted Autogenic Drainage (AAD) or bouncing combined with Assisted Autogenic Drainage (BAAD), induces or aggravates acid and non-acid gastro-oesophageal reflux in infants under the age of one year. Infants, referred to the hospital for impedance-pH monitoring are included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Each child under the age of 1 year, referred for 24 h impedance monitoring to confirm a clinically suspected diagnosis of pathological GOR will be included

Exclusion Criteria:

* prematurity (gestational age less than 37 weeks),
* the use of anti-reflux medication and reflux surgery (Nissen fundoplication)

Ages: 1 Day to 365 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
number of refluxes | 20 minutes

SECONDARY OUTCOMES:
number of acid refluxes | 20 minutes

OTHER OUTCOMES:
number of non-acid refluxes | 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Filip Van Ginderdeuren, PhD, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- UZBrussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No